CLINICAL TRIAL: NCT04831190
Title: ACE-Neuro: A Tailored Exercise Oncology Program for Neuro-Oncology Patients
Brief Title: A Tailored Exercise Oncology Program for Neuro-Oncology Patients
Acronym: ACE-Neuro
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Collaborators: Alberta Cancer Foundation (Other); University of Alberta (Other); Tom Baker Cancer Centre (Other); Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-20-0322
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Cancer; Brain Tumor, Primary
Keywords: Neuro-Oncology; Cancer; Exercise; Quality of Life; Feasibility; Implementation
MeSH Terms: conditions — Neoplasms; Brain Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Feasibility-Implementation Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All participants will be involved in a tailored exercise intervention for 12 weeks.
  Interventions: Behavioral: Tailored Exercise Intervention

INTERVENTIONS:
Behavioral: Tailored Exercise Intervention — The exercise program to be implemented for neuro-oncology patients will combine aerobic, resistance, balance, and flexibility exercises delivered in one-to-one setting (i.e., personal training) twice per week, for 12 weeks. Based on needs and preferences, participants will have the option to join a circuit-type group class once per week in place of one of their personal training sessions. During COVID-19, all sessions will be delivered remotely. If facilities are open and deemed safe for cancer patients, participants will have the option to attend an in-person session, integrated in the community. Whether delivered in-class or remotely, the intervention will follow exercise progression principles (i.e., frequency, intensity, time, type, overload, and progression) over the 12-weeks, with tailoring of any exercise to meet individual participant needs, with aims of promoting wellness and physical function. The exercise intervention is based on the Alberta Cancer Exercise (ACE) program.

SUMMARY:
Background: Exercise, or physical activity, is beneficial for all cancer survivors. Despite this knowledge, there is generally a gap between the evidence and practice. And this gap is widened with (a) underserved tumour groups in exercise oncology, such as neuro-oncology patients, or (b) underutilized timelines across the cancer treatment phases to deliver exercise oncology education or programming. Thus, our current work is building a hybrid implementation effectiveness study into the clinical care pathway across Alberta in neuro-oncology - ACE-Neuro.

Objectives: The purpose of this study is to assess the impact of an online, tailored exercise oncology program for neuro-oncology patients using a participant-oriented research (POR) approach as well as both quantitative and qualitative research methods. Specifically, the primary outcome of this study is to determine the feasibility of recruitment, referral, triage, adherence, and adverse events. The secondary outcome is to examine the preliminary effectiveness of the neuro-oncology exercise program on patient-reported outcomes and physical function.

Methods: Neuro-oncology patients >18 years and able to consent in English will be referred to a study-based Rehabilitation Triage Clinic, where a Physician-Researcher will assess patients on their overall health and functional status, and next triage them to either ACE-Neuro, rehabilitation oncology, or cancer physiatry. Once referred to ACE-Neuro, participants will partake in a 12-week online exercise program, delivered by a Clinical Exercise Physiologist. Participants will complete online assessments of physical function, patient-reported outcomes, and objective physical activity at baseline (pre-program), 12-weeks (post-program completion), 6-months, and 12-months. The exercise program includes weekly one-on-one online exercise delivery, health coaching to support behaviour change, and access to an online group exercise session. Participants will also be invited to a post-program qualitative interview to get perspectives on their experiences participating in ACE-Neuro.

Relevance: By working directly with patients, healthcare providers, and community partners, this implementation project will develop a framework that streamlines patient triage, and provides a tailored online exercise program for neuro-oncology patients, thereby advancing exercise oncology research and clinical practice.

DETAILED DESCRIPTION:
BACKGROUND & RATIONALE

Exercise, or physical activity, is beneficial for all cancer survivors. Despite this knowledge, there is generally a gap between the evidence and practice. And this gap is widened with (a) underserved tumour groups in exercise oncology, such as neuro-oncology patients, or (b) underutilized timelines across the cancer treatment phases to deliver exercise oncology education or programming.

Within Alberta (AB), the investigators have been able to very successfully implement the Alberta Cancer Exercise (ACE) program to start to address the gap between research and practice. As a hybrid implementation effectiveness study, ACE is building a model for exercise oncology delivery within standard cancer care. With over 2500 participants across AB, the investigators have substantial evidence supporting the feasibility of ACE, as well as the potential benefits. Despite these successes, ACE remains primarily represented by participants from breast, prostate, and colorectal tumour groups. This represents a lack of connection between smaller and more high risk tumour groups within referral pathways for the ACE program, both at TBCC and CCI, but also within the regional community cancer clinics (Grande Prairie, Red Deer, Medicine Hat, Lethbridge).

RESEARCH QUESTION & OBJECTIVES

The purpose of this feasibility-implementation study is to build exercise into the clinical care pathway in neuro-oncology clinics at the two major cancer centres in AB, where all neuro-oncology patients provincially are treated (Tom Baker Cancer Centre, TBCC; and the Cross Cancer Institute, CCI). Specifically, the objectives of the proposed work are: (1) to tailor the ACE exercise program for all neuro- oncology patients, to ACE-Neuro; this includes considering additional tailoring to address needs earlier in the care pathway, from diagnosis through treatment (i.e., prehabilitation phases) and into longer term survivorship (wellness cancer survivorship care plans), (2) to provide models of delivery of exercise oncology programs to enhance access (i.e., remote delivery, home support, individual vs group), and (3) to build this systematically within the neuro-oncology clinics at the TBCC and CCI, to ensure that all patients diagnosed with brain tumours can access wellness during their cancer care journey. The investigators hypothesize that there will be improvements in patients' physical and psychosocial well-being (individual level outcomes), as well as a more integrated workflow in the clinical cancer care setting that includes exercise as part of standard clinical practice (systems level outcome). Specifically, the primary outcome of this study is to determine the feasibility of recruitment, referral, triage, adherence, and adverse events. The secondary outcome is to examine the preliminary effectiveness of the neuro-oncology exercise program on patient-reported outcomes and physical function.

METHODS

Using the successful implementation model developed in ACE, the proposed work will build a neuro-oncology cohort within a mixed methods study design. There will be multiple phases to the implementation of ACE-Neuro, including:

1. Building awareness within the clinical teams, identifying site champions, and providing educational and referral resources specific to neuro-oncology and exercise;
2. Working with neuro-oncology patients and families to develop the unique aspects of exercise programming (from "move more" programs to "exercise") to address identified needs. This co-creation process will also include the cancer physiatry team (Dr. George Francis, Dr. Lauren Capozzi) and the clinical neuro-oncology teams (Dr. Gloria Roldan Urgoiti at TBCC and Dr. Jay Easaw at CCI) to address medical clinical needs that can be addressed within the ACE-Neuro program, and clinical workflow logistics with physiatry and physiotherapy to address specific treatment-related side effects (such as limb weakness, balance, or cognitive function);
3. implementation of the ACE-Neuro tailored program, including referral, screening, assessments, intervention delivery, and follow-ups. Details of the ACE-Neuro procedures are detailed below.

REFERRAL AND RECRUITMENT

Because the main outcome of this study is feasibility, and the ultimate goal is to build ACE-Neuro into standard neuro-oncology care, no a priori sample size has been calculated. Based on current clinical numbers, and previous work done with neuro-oncology patients at CCI, the investigators anticipate approximately 25-30 eligible patients per year, per site. Our aim is to referral of all eligible neuro-oncology patients from TBCC. For recruitment, patients can:

1. self-refer (i.e. patient contacts the study team from a poster or brochure received in clinic, through word of mouth);

   OR study team can refer:
2. clinical team sends referral to rehab oncology via Putting Patients First Questionnaire (via ARIA).

The clinical team, based on their judgment, may not refer patients they deem to be ineligible. This may include for the following reasons:

1. Patient is not interested when exercise idea is brought up.
2. Health care provider deems patient clinically ineligible, due to disease progression, end-of-life care, or other health factor
3. Patient does not speak English
4. Other

As a feasibility study, reasons for non-referral will be tracked, with no identifying patient information, across the recruitment period. After consenting to the study, all patients will undergo a two-part screening procedure prior to beginning the exercise program:

1. Patients will complete health and medical history screening using the Health History Questionnaire, Identifying Information Questionnaire, and the Physical Activity Readiness Questionnaire; PAR-Q.
2. Patients will attend a Neuro Oncology Rehabilitation Triage Clinic, led by a Resident Physician (Dr. Lauren Capozzi; supervised by Dr. George Francis) and the ACE-Neuro Study Coordinator (Julia Daun). During this 30-minute appointment, patients will complete the Short Physical Performance Battery screening test6, and a full neurological exam, including Karnofsky performance and Eastern Cooperative Oncology Group (ECOG) scores. This appointment will assess the patients' readiness for participating in ACE-Neuro.

As part of this study, the investigators will be tracking the referral pathway, and which method of referral is most feasible as part of standard clinical workflow.

ASSESSMENTS

1. Patient-Reported Outcomes (PROs) - will include symptom burden (Edmonton Symptom Assessment Scale-Revised; ESAS-r), PA levels (Godin Leisure Time Exercise Questionnaire-Modified; GLTEQ), quality of life (Functional Assessment of Cancer Therapy-Brain; FACT-Br), cognitive function (Functional Assessment of Cancer Therapy-Cognitive Scale; FACT-Cog), and fatigue (Functional Assessment of Chronic Illness Therapy-Fatigue; FACIT-F).
2. Functional Fitness Assessments - will follow the set protocols within ACE (HREBA-CC-16- 0905_MOD12), and are designed to be able to be completed in-person or via remote delivery (online assessment). All fitness assessments will be completed by a Clinical Exercise Physiologist and will include the assessment of lower body strength and endurance (30-second sit-to-stand), static balance (single leg stance), flexibility (sit-and-reach and active shoulder flexion), and cardiorespiratory fitness (2-minute step test or 6MWT).
3. Objective Physical Activity - will be measured via the use of a wrist-worn activity tracker (WAT; i.e., Garmin vivosmart® 4). Garmin wearable PA trackers are widely used across health research, and will be provided to all participants to objectively track PA habits throughout the intervention.
4. Qualitative Interviews and Photo Elicitation: Qualitative data will be gathered across the co-creation process via interviews and photo elicitation, to inform the feasibility of ACE-Neuro, as well as to assess outcomes associated with participation in the ACE-Neuro program (benefits, barriers, satisfaction, impact on well-being). Qualitative data will be stored on a secure server.

HEALTH COACHING

In addition to exercise delivery and assessments, all participants will have the choice to participate in evidence-based health coaching calls, provided by a trained Health Coach. Health coaching is an evidence-based tool that supports positive health behaviour change across cancer populations. Health coaching calls will take place weekly for 15-30 minutes following an individualized exercise training session, and include topics surrounding goal setting, social support, stress management, maintaining motivation, and overcoming barriers. Health coaching calls will be delivered remotely (e.g., via end-to-end encrypted Zoom or phone call) at the participants' preferred date and time.

TIMELINE

The described exercise program and data collection of PROs and functional fitness assessments are in addition to standard practices. The timeline for these assessments include: baseline (at recruitment into ACE-Neuro), 12-weeks (post-intervention), 6-months, and 12-months.

ANALYSIS Quantitative analysis will include descriptive statistics (means, medians, standard deviations), and change scores to measure changes in outcomes over time. Qualitative data will be analyzed by verbatim transcription (in NVivo), using an interpretive description methodology. Both quantitative and qualitative data will be analyzed to provide a deeper understanding of the feasibility and impact of ACE-Neuro.

RELEVANCE By working directly with patients, healthcare providers, and community partners, this implementation project will develop a framework that streamlines patient triage, and provides a tailored online exercise program for neuro-oncology patients, thereby advancing exercise oncology research and clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* are a neuro-oncology patient with primary brain tumour (malignant or benign)
* are pre-, on, or completed treatment
* are over the age of 18 years
* are able to read/write in English
* are able to participate in mild levels of exercise
* are able to access remote programming (i.e., has internet access and a computer or tablet)

Exclusion Criteria:

* diagnosis is not primary brain
* unable to read/write in English
* are unable to participate in light exercise
* for online programs, do not have internet or computer access

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Referral: Referral Rate | From start of study recruitment to end of study (2 years).
  The percentage of patient referrals to the study team from the clinical team from patients eligible.
Feasibility of Enrolment: Enrolment Rate | From start of study recruitment to end of study (2 years).
  The percentage of patients that enrol in the study once they hear the full study introduction.
Feasibility of Triage: Triage Completion Rate | From start of study recruitment to end of study (2 years).
  The percentage of participants that attend, from those that are referred, to the Neuro-Oncology Rehabilitation Triage Clinic.
Feasibility of Program Attendance: Program Attendance Rate | Baseline to 12 weeks.
  Percentage of classes attended by enrolled participants.
Feasibility of Measurement Completion: Measurement Completion Rate (Baseline) | At baseline (0 weeks).
  Percentage of measures (i.e., patient-reported outcomes and physical function) completed by enrolled participants.
Feasibility of Measurement Completion: Measurement Completion Rate (12 Weeks) | Post-program completion (12 weeks).
  Percentage of measures (i.e., patient-reported outcomes and physical function) completed by enrolled participants.
Feasibility of Measurement Completion: Measurement Completion Rate (6 Months) | At 6 months post study enrolment.
  Percentage of measures (i.e., patient-reported outcomes and physical function) completed by enrolled participants.
Feasibility of Measurement Completion: Measurement Completion Rate (12 Months) | At 12 months post study enrolment.
  Percentage of measures (i.e., patient-reported outcomes and physical function) completed by enrolled participants.
Safety of Intervention | Baseline to 12 weeks.
  Record of any adverse events related to the intervention.
Attrition Rate | Baseline to 12 weeks.
  Number of participants who consent but do not complete the intervention.
Qualitative Feasibility: Qualitative Semi-Structured One-on-One Interviews | Conducted between weeks 12-14.
  Participant perception of intervention feasibility via semi-structured one-on-one interviews (qualitative data, not reported on a scale).

SECONDARY OUTCOMES:
Physical Activity Minutes Per Week | Baseline to 12 weeks.
  Change in number of participants meeting Guidelines for Physical Activity of 90 minutes per week of moderate intensity exercise, based on accelerometer data from commercially-available activity tracker (Garmin vivosmart® 4).
Weekly Step Count | Baseline to 12 weeks.
  Total weekly step count based on data from commercially-available activity tracker (Garmin vivosmart® 4).
Body Composition | Baseline to post 12-week exercise intervention.
  Measure of change in body mass index (BMI) over time.
Cardiorespiratory Fitness | Baseline to post 12-week exercise intervention and maintenance of change from 12-weeks to 6-months; and from 12 weeks to 12 months.
  Change in 6-minute walk test (m) or 2-minute step test (steps) results.
Muscular Strength | Baseline to post 12-week exercise intervention and maintenance of change from 12-weeks to 6-months; and from 12 weeks to 12 months.
  Change in hand-grip dynamometry (kg).
Muscular Endurance | Baseline to post 12-week exercise intervention and maintenance of change from 12-weeks to 6-months; and from 12 weeks to 12 months.
  Change in sit-to-stand (number of repetitions in 30 seconds).
Upper Extremity Flexibility | Baseline to post 12-week exercise intervention and maintenance of change from 12-weeks to 6-months; and from 12 weeks to 12 months.
  Change in active shoulder flexion range of motion (degrees).
Lower Extremity Flexibility | Baseline to post 12-week exercise intervention and maintenance of change from 12-weeks to 6-months; and from 12 weeks to 12 months.
  Change in sit-and-reach test (cm).
Static Balance | Baseline to post 12-week exercise intervention and maintenance of change from 12-weeks to 6-months; and from 12 weeks to 12 months.
  Change in one single-leg-stance test (seconds).
Symptom Burden | Baseline to post 12-week exercise intervention and maintenance of change from 12-weeks to 6-months; and from 12 weeks to 12 months.
  Change in Edmonton Symptom Assessment Scale. Scale includes 10 questions total and is from 0-10, where 0 means the symptom is absent and 10 means the worst possible severity of the symptom is being experienced. Total score 0-100, higher is worse.
Subjective Reporting of Average Weekly Physical Activity | Baseline to post 12-week exercise intervention and maintenance of change from 12-weeks to 6-months; and from 12 weeks to 12 months.
  Change in Godin Leisure Time Exercise Questionnaire (GLTEQ). Self-reported as total minutes of physical activity in the past week. Calculated as [mild frequency per week x 3] + [moderate frequency per week x 5] + [strenuous frequency per week x 9]. Minimum score is 0, the maximum is dependent on the participant's frequency of physical activity. Higher score indicates more physical activity.
Fatigue | Baseline to post 12-week exercise intervention and maintenance of change from 12-weeks to 6-months; and from 12 weeks to 12 months.
  Change in Functional Assessment of Chronic Illness Therapy - Fatigue subscale Scale is from 0-4, where 0 means "not at all" and 4 means "very much". Total score 0-52, higher score is lower fatigue severity.
Quality of Life - Brain Subscale | Baseline to post 12-week exercise intervention and maintenance of change from 12-weeks to 6-months; and from 12 weeks to 12 months.
  Change in Functional Assessment of Cancer Therapy - Brain Subscale. Scale is from 0-4, where 0 means "not at all" and 4 means "very much". Total score ranges from 0-200. A higher score indicates a better outcome.
Cognition | Baseline to post 12-week exercise intervention and maintenance of change from 12-weeks to 6-months; and from 12 weeks to 12 months.
  Change in Functional Assessment of Cancer Therapy - Cognitive Subscale. Scale is from 0-4, where 0 means "never" and 4 means "several times a day" (experiencing symptoms). Total score ranges from 0-80. A higher score indicates a better outcome.
Program Implementation and Evaluation | Baseline to 2 years.
  The RE-AIM Framework: program reach, effectiveness, adoption, implementation and maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: S. Nicole Culos-Reed, PhD, Principal Investigator — University of Calgary, Calgary, AB, Canada; Gloria Roldan Urgoiti, MD, Principal Investigator — Department of Medical Oncology, Tom Baker Cancer Centre, Calgary, AB, Canada; Jay Easaw, MD, Principal Investigator — Department of Oncology, Cross Cancer Institute, Edmonton, AB, Canada; Margaret McNeely, PT, PhD, Principal Investigator — University of Alberta, Edmonton, AB, Canada
Locations (4):
- Canada (4):
  - Health and Wellness Lab, University of Calgary, Calgary, Alberta
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, University of Alberta, Edmonton, Alberta
  - Cancer Rehabilitation Clinic, Faculty of Rehabilitation Medicine, University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No
No plan at this time to share IPD outside of the research team.

REFERENCES:
- [Derived] Daun JT, Capozzi LC, Dhruva T, Roldan Urgoiti G, McDonough MH, McLaughlin E, Bansal M, Brett A, Easaw JC, McNeely ML, Francis GJ, Williamson T, Danyluk J, Ospina PA, Lesiuk C, de Robles P, Leckie C, Culos-Reed SN. The feasibility of a multi-site, clinic-supported, and tailored neuro-oncology exercise program. Neurooncol Pract. 2024 Oct 10;12(1):131-142. doi: 10.1093/nop/npae093. eCollection 2025 Feb. PMID 39917754